CLINICAL TRIAL: NCT00363519
Title: MK-0431/ONO-5435 Phase III Clinical Study - Glimepiride add-on Study for Patients With Type 2 Diabetes Mellitus
Brief Title: Controlled Study of MK-0431/ONO-5435 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ONO-5435-09
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MK-0431; ONO-5435; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- P (Placebo Comparator)
  Interventions: Drug: Placebo
- E (Experimental)
  Interventions: Drug: Sitagliptin phosphate

INTERVENTIONS:
Drug: Placebo — Double-blind period (12 wk); placebo QD The double-blind period will be followed by a 40 wk open-label extension period where MK-0431/ONO-5435 could be titrated from 50 mg QD to 100 mg QD
  Arms: P
Drug: Sitagliptin phosphate — Double-blind period (12 wk); 50 mg QD The double-blind period will be followed by a 40 wk open-label extension period where MK-0431/ONO-5435 could be titrated from 50 mg QD to 100 mg QD
  Arms: E

SUMMARY:
The purpose of this study is to determine the safety and efficacy of MK-0431/ONO-5435 in patients with Type 2 diabetes mellitus who have inadequate glycemic control on diet/exercise therapy and glimepiride as monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus on diet/exercise therapy and glimepiride as monotherapy

Exclusion Criteria:

* Patients with Type 1 diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
safety | 52 weeks
tolerability | 52 weeks

SECONDARY OUTCOMES:
Plasma glucose | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikio Nishii, Study Director — Ono Pharmaceutical Co. Ltd
Locations (8):
- Japan (8):
  - Chugoku Region, Chugoku
  - Chubu Region, Chūbu
  - Hokkaido Region, Hokkaido
  - Kanto Region, Kanto
  - Kinki Region, Kinki
  - Kyushu Region, Kyushu
  - Shikoku Region, Shikoku
  - Tohoku Region, Tōhoku